CLINICAL TRIAL: NCT03657511
Title: Educational Interventions to Promote Tobacco Cessation Among Women Seeking Mammography Screening
Brief Title: Tobacco Cessation Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Responsible Party: Principal Investigator, Ann Schwartz, Principal Investigator, Barbara Ann Karmanos Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2018-006
Record Dates: First submitted 2018-08-31; First posted 2018-09-05 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2022-05

CONDITIONS: Smoking Tobacco
Keywords: Smoking
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Educational Interventions to Promote Tobacco Cessation (Other)
  Interventions: Behavioral: Educational Interventions to Promote Tobacco Cessation

INTERVENTIONS:
Behavioral: Educational Interventions to Promote Tobacco Cessation — Women receiving a screening mammogram at KCI downtown and McLaren Macomb, will be given a self-administered questionnaire at check-in.
  Women who indicate they are current smokers are eligible for the study. After the screening mammogram is complete, eligible women will be consented. Educational materials will be provided to the participant at that time. The materials provided outline evidence-based approaches to smoking cessation and include contact information for local resources including cessation support groups, Michigan Tobacco Quitline, American Cancer Society's Guide to Quitting Smoking, Quitnet, Smokfree.gov and Become An Ex. The participant will be contacted by telephone approximately 12 weeks later to determine if she is currently smoking or had quit in the last 12 weeks.

SUMMARY:
This study is planned as an evaluation of a low cost, simple smoking cessation intervention. There is very little information about the effectiveness of a simple tobacco cessation strategy. Therefore, our objective is to obtain estimates of effectiveness that can be used to refine existing programs or to develop new ones.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and read English

Exclusion Criteria:

* Currently undergoing tobacco cessation treatment

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 100 (Actual)
Dates: Start 2018-10-22 (Actual); Primary Completion 2021-06-21 (Actual); Study Completion 2021-06-21 (Actual)

PRIMARY OUTCOMES:
The number of women who quit smoking in the last 12 weeks | 12 weeks after initial self-administered questionnaire
  Completion of second questionnaire to determine if participant is currently smoking or had quit smoking in the last 12 weeks.

SECONDARY OUTCOMES:
The number of women who attempted to quit smoking in the last 12 weeks. | 12 weeks after initial self-administered questionnaire
  Completion of second questionnaire to determine if participant is currently smoking or had quit smoking in the last 12 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- Barbara Ann Karmanos Cancer Institute, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No